CLINICAL TRIAL: NCT03270605
Title: Myomectomy During Cesarean Section: A Retrospective Cohort Study
Brief Title: Myomectomy During CS: A Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: R/17.04.71
Record Dates: First submitted 2017-08-31; First posted 2017-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Cesarean Section; Uterine Fibroid
MeSH Terms: conditions — Leiomyoma | interventions — Uterine Myomectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CS with myomectomy: Women having uterine myoma with pregnancy and subjected to myomectomy during delivery by CS
  Interventions: Procedure: Myomectomy
- CS without myomectomy: Women having uterine myoma with pregnancy and delivered by CS without myomectomy

INTERVENTIONS:
Procedure: Myomectomy — Surgical removal of uterine fibroid
  Groups: CS with myomectomy

SUMMARY:
To evaluate the value of myomectomy during delivery by cesarean section (CS) in pregnant women with uterine fibroids.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent elective CS with presence of uterine fibroid during the index pregnancy documented antenatal and at surgery

Exclusion Criteria:

* Antepartum hemorrhage
* Blood diseases or bleeding tendencies.
* Medical conditions complicating pregnancy.
* Performed another surgical procedure at CS other than myomectomy.

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with uterine fibroid during the index pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Deficit in hemoglobin level | 24 hours
  Preoperative hemoglobin minus postoperative hemoglobin level (in gm/dl)

SECONDARY OUTCOMES:
Operative time | 3 hours
  Time to complete the procedure
Postoperative hospital stay period | 7 days
  Time from the end of operation to discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Waleed El-refaie, MD, Principal Investigator — Port Said University; Mohamed Hassan, MD, Study Director — Mansoura University; Mohamed S Abdelhafez, MD, Study Chair — Mansoura University

IPD SHARING:
Plan to Share IPD: Undecided